CLINICAL TRIAL: NCT06762652
Title: ImpRovEd Care After eSophageCtomy Using an Algorithm for postoperativE Complications - RESCUE Trial
Acronym: RESCUE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other); Erasmus Medical Center (Other); University Medical Center Groningen (Other); Hospital Group Twente (ZGT) (Unknown); Antoni van Leeuwenhoek Hospital (Other); Leiden University Medical Center (Other); Elisabeth-TweeSteden Ziekenhuis (Other); medical center leeuwarden (Unknown); Zuyderland Medical Centre (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Reinier de Graaf Groep (Other); Gelre Hospitals (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024-17562; 10390032310024 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-12-19; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Diagnosis and Treatment of Complications After Esophagectomy
Keywords: diagnosis; treatment; complications; esophagectomy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized superiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual Care (Active Comparator): During the control period, (participating) patients will receive usual postoperative care. Postoperative care, including diagnosis and management of postoperative complications, will be performed in line with local standards and/or protocols. For diagnosis of complications, physicians may perform laboratory tests such as CRP or leucocyte count, and diagnostic imaging such as CT-scan, X-ray or endoscopy. For treatment of complications, conservative, radiological, endoscopic and surgical treatments are often applied.
  Interventions: Other: Wash-in period; Diagnostic Test: Algorithm-based care

INTERVENTIONS:
Other: Wash-in period — The goal of the wash-in period between the control and intervention period is to intensively educate and train physicians to use the algorithm as intended during daily postoperative care. The coordinating investigator along with the local principal investigator will be responsible for this training. Training will be performed in a standardized approach in order to guarantee uniformity across centres.
Diagnostic Test: Algorithm-based care — During the intervention period, (participating) patients will receive algorithm-based care. The RESCUE algorithm is a consensus-based clinical care algorithm developed to standardize postoperative care. The algorithm includes the same modalities as applied in usual care, and does not include novel/experimental modalities, but rather offers a novel, standardized approach to guide the use of common modalities during postoperative care. The daily objective evaluation of patients' condition, vital signs and biochemical parameters is thought to aid early diagnosis of complications after esophagectomy which enables treatment before systemic symptoms become apparent and prevent development of sepsis. Physicians are always allowed to deviate from the RESCUE, but reasons for deviating will be recorded.

SUMMARY:
The objective of the RESCUE-trial is to investigate whether implementation of a consensus-based clinical care algorithm to standardize diagnosis and management of postoperative complications reduces 90-day mortality, ICU (re)admission and surgical interventions after esophagectomy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Age ≥ 18 years
2. Histologically proven esophageal or gastro-esophageal junction carcinoma (cT1-4aN0-3M0)
3. Scheduled to undergo curatively-intended esophagectomy with gastric tube reconstruction. All techniques (i.e. minimally invasive, robotic, hybrid, open) and approaches (i.e. transthoracic, transcervical, transhiatal) of esophagectomy are suitable for inclusion.
4. Ability to provide written informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Emergency resection
2. Patients who underwent (additional) total gastrectomy
3. Patients who underwent reconstruction using colonic or jejunal interposition
4. Patients in whom no anastomosis is created during resection
5. Secondary malignancy which determines prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Severe complications | 90 days
  The primary outcome measure is the incidence of severe complications (i.e. Clavien-Dindo ≥ 3b). Severe complications are defined as a composite endpoint with one or more of the following criteria within 90 days after esophagectomy:
  1. The complication was treated under general anaesthesia.
  2. Postoperative mortality.
  3. Escalation of care due to new onset or progressive organ failure (i.e. patients requiring vasopression, dialysis, (re-)intubation, (re)admission to a medium care or intensive care unit).

SECONDARY OUTCOMES:
General quality of life | 6 weeks, and 3, 6, and 12 months after esophagectomy
  General quality of life, as measured using the validated EuroQol EQ-5D-5L questionnaire. Assessment will be performed at 6 weeks and 3, 6 and 12 months.
Time to functional recovery | 90 days after esophagectomy
  Time to functional recovery, defined as when a patient does not need intravenous fluid, has adequate pain control with oral analgesia (Numeric Rating Scale ≤4), restored mobility to an independent level (e.g. walk to the toilet with(out) walking aids and transfer bed/chair) or back to the previous functioning level of mobilization, sufficient caloric intake (minimum of 50% of the required calories), no signs of an active infection (no fever and declining CRP levels).
Comprehensive Complications index | 90 days after esophagectomy
  Comprehensive Complications Index, a measure for the severity of all complications together.
Failure to rescue | 90 days after esophagectomy
  Failure to rescue, defined as the rate of mortality in patients with a complication within 90-days after esophagectomy.
Length of hospital (intensive care unit) stay | 90 days after esophagectomy
  Length of hospital and ICU stay, defined as the amount of days the patient stays in the ICU and in the hospital during 90 days postoperatively.
Succes of algorithm implementation | 90 days after esophagectomy
  succes of implementation (i.e. proportion of patients' days in which the algorithm was not followed)
Economic evaluation | 3,6 and 12 months after esophagectomy
  Cost-efficacy analysis will be performed from a societal perspective, including both medical and non-medical costs. Economic evaluation will be performed at 12 months follow-up. Medical resource use will be recorded from hospital records, including length of stay, laboratory and diagnostics use and treatment of complications. Medical resource use as well as out-of-pocket expenses will be recorded using iMTA Medical Consumption Questionnaire (iMCQ). [26] Resource use will be multiplied by associated unit costs to obtain total costs. Standard cost prices from the 'Dutch Guidelines for Cost Analyses' and www.medicijnkosten.nl will be used. Volumes of care will be multiplied by the cost price of each volume to calculate costs.
Productivity losses | 3,6 and 12 months after esophagectomy
  Productivity losses will be measured using the iMTA Productivity Cost Questionnaire (iPCQ).
Budget Impact Analysis | 3,6 and 12 months after esophagectomy
  Budget Impact Analysis (BIA) will be performed to assess the financial consequences of implementing the algorithm-based care, wherein the internationally accepted principles of ISPOR for the design, implementation and reporting of the BIA will be used. The third party payer perspective will be adopted to inform a business case for reimbursement companies.
Cancer-specific quality of life | 6 weeks, and 3, 6, and 12 months after esophagectomy
  Cancer-specific quality of life, as measured using the validated EIRTC QLQ-C30 questionnaire. Assessment will be performed at 6 weeks and 3, 6 and 12 months.
Esophageal cancer-specific quality of life | 6 weeks, and 3, 6, and 12 months after esophagectomy
  Esophageal cancer-specific quality of life, as measured using the validated EORTC QLQ-OG25 questionnaire. Assessment will be performed at 6 weeks and 3, 6 and 12 months.

IPD SHARING:
Plan to Share IPD: Undecided
This concerns a conceptual registration.